CLINICAL TRIAL: NCT04171999
Title: CommunityRx-Hunger: A Hospital-based Intervention for Primary Caregivers of Children Admitted to the Hospital
Brief Title: CommunityRx-Hunger
Acronym: CRx-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB20-0324; 1R01MD012630-01A1 (NIH)
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2023-11

CONDITIONS: Food Insecurity
Keywords: Food Insecurity; Caregivers; Clinical Trial; Hunger; Self-Efficacy; Health-Related Social Needs

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-Blind randomized controlled trial where the data collectors are blinded to the condition to which the subject has been assigned. The subject is also blinded to the condition they are assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care + Intervention (Case) (Experimental): Cases will receive the CommunityRx Intervention.
  Interventions: Other: Community Rx-Hunger (CRx-H)
- Usual Care (Control) (No Intervention): Controls will receive the usual standard care, which consists of information about hospital food resources and access to Feed1st hospital food pantries prior to discharge.

INTERVENTIONS:
Other: Community Rx-Hunger (CRx-H) — The CRx-H Intervention provides "dosages" of health content that offer assistance for food insecurity and other health-related social needs. A caregiver randomized to the intervention will receive a hard-copy print-out of their tailored list of resources to address food insecurity. A member of our research team will deliver this list and provide a brief educational component which includes: a brief, structured script about the common problem of food insecurity in households with children and co-occuring HRSNs, review of the resource list which includes nearby, vetted resources to address these needs and coaching on how to activate resources on the list. Prior to discharge, the caregiver will receive a duplicate copy of the list of resources. After discharge, the caregiver will receive text messages at a frequency based on the Critical Time Intervention (CTI) Model, from baseline to 3 months post discharge, in order to receive ongoing support by a research team member.
  Arms: Usual Care + Intervention (Case)

SUMMARY:
CommunityRx-Hunger (CRx-H) is a hospital-based intervention that addresses food insecurity and other health-related social needs such as transportation, housing, utilities, and safety. Study team members are recruiting caregivers at the time of their child's hospital admission at a large urban children's hospital. For Aim 1, the primary outcome is self-efficacy among food insecure caregivers compared to those who receive the usual standard of care. For Aim 2, the primary outcome is satisfaction with care compared between food secure and food insecure caregivers.

DETAILED DESCRIPTION:
CommunityRx-Hunger (CRx-H) is a double-blinded randomized controlled trial aimed at increasing self-efficacy among caregivers with food insecurity in the household. CRx-H is recruiting primary caregivers of hospitalized children at a large urban children's hospital at the time of admission. Aim 1: Researchers are studying whether the intervention will increase self-efficacy among food insecure caregivers compared to those who receive the usual standard of care. Aim 2: Researchers will enroll and randomize caregivers with and without food insecurity to the intervention to compare satisfaction with care.

Eligible, self-identified caregivers will complete a baseline survey during the child's hospital stay, followed by phone surveys at 7, 30, 90, 180 days, and 12 months. Caregivers randomized to the intervention will receive a tailored list of resources to address food insecurity and other health-related social needs, plus a brief educational component delivered by a trained member of our research team. Cases will receive a "booster" dose of the resource list prior to discharge. After discharge, cases will receive proactive text messages about those same community resources.

All caregivers (regardless of research arm) will receive a series of text messages related to the study such as reminders to schedule the phone survey with a member of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Native English or Spanish speaker
* Living in 1 of 27 zip codes in the study's target region
* Self-identify as a primary caregiver of a child <18 years old hospitalized in a large urban children's hospital
* Ability to send and receive text messages
* Access to a mobile phone and agrees to receive text messages from the study

Exclusion Criteria:

* Previous participation in a CRx research study.
* Caregivers of newborns in the hospital
* Patient hospital stay is less than 24 hours
* Patient hospital stay is 30 days or more
* Patient has an eating disorder as indicated in the EMR

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy T Lindau, MD, MPP, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Lindau ST, Makelarski JA, Winslow VA, Abramsohn EM, Anand V, Burnet DL, Fuller CM, Grana M, Miller DC, Ren ES, Waxman E, Wroblewski KE. Low-Intensity Social Care and Child Acute Health Care Utilization: A Randomized Clinical Trial. JAMA Pediatr. 2025 Jun 1;179(6):610-620. doi: 10.1001/jamapediatrics.2025.0484. PMID 40293738
- [Derived] Glasser NJ, Lindau ST, Wroblewski K, Abramsohn EM, Burnet DL, Fuller CM, Miller DC, O'Malley CA, Shiu E, Waxman E, Makelarski JA; CommunityRx-Hunger Collaborators. Effect of a Social Care Intervention on Health Care Experiences of Caregivers of Hospitalized Children: A Randomized Clinical Trial. JAMA Pediatr. 2023 Dec 1;177(12):1266-1275. doi: 10.1001/jamapediatrics.2023.4596. PMID 37902777
- [Derived] Abramsohn EM, De Ornelas M, Borson S, Frazier CRM, Fuller CM, Grana M, Huang ES, Jagai JS, Makelarski JA, Miller D, Schulman-Green D, Shiu E, Thompson K, Winslow V, Wroblewski K, Lindau ST. CommunityRx, a social care assistance intervention for family and friend caregivers delivered at the point of care: two concurrent blinded randomized controlled trials. Trials. 2023 Oct 21;24(1):681. doi: 10.1186/s13063-023-07697-z. PMID 37864258
- [Derived] Abramsohn EM, De Ornelas M, Borson S, Frazier CR, Fuller CM, Grana M, Huang ES, Jagai JS, Makelarski JA, Miller D, Schulman-Green D, Shiu E, Thompson K, Winslow V, Wroblewski K, Lindau ST. Two concurrent randomized controlled trials of CommunityRx, a social care intervention for family and friend caregivers delivered at the point of care. Res Sq [Preprint]. 2023 Mar 1:rs.3.rs-2464681. doi: 10.21203/rs.3.rs-2464681/v1. PMID 36909590

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to the randomized trial, 20 participants were enrolled as part of pre-testing.
Period: Overall Study
Arm/Group | Usual Care + Intervention (Case) | Usual Care (Control)
Started | 320 | 320
Completed | 318 | 319
Not Completed | 2 | 1
Not completed — deemed ineligible after randomization | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care + Intervention (Case) | Usual Care (Control) | Total
Number analyzed (Participants) | 318 | 319 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (9.2) | 34.9 (9.2) | 35 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall due to missing data and other response.
  Participants
    number analyzed (Participants) | 316 | 319 | 635
    Female | 298 | 302 | 600
    Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 41 | 92
  Not Hispanic or Latino | 267 | 278 | 545
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 246 | 259 | 505
  White | 36 | 27 | 63
  More than one race | 6 | 12 | 18
  Other | 25 | 19 | 44
  Unknown or not reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: (Aim 1) Caregiver Self-efficacy at 12 Months Among Food Insecure Caregivers
Description: Self-efficacy is measured by Bandura's Self-Efficacy Scale which asks, "How confident are you in your ability to find resources in your community that help you manage your health?" Responses will be assessed on a 5-point Likert scale ranging from "not at all confident" to "completely confident."
Time Frame: 12 months
Population: Analysis was restricted to caregivers who were food insecure at baseline and who completed the self-efficacy measure at 12 month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care + Intervention (Case) | Usual Care (Control)
Number analyzed (Participants) | 74 | 74
Participants
  Not at all confident | 2 | 5
  Not very confident | 9 | 4
  Uncertain | 13 | 6
  Somewhat confident | 18 | 33
  Completely confident | 32 | 26

2. Primary Outcome: (Aim 2) Caregiver Satisfaction With Hospital Discharge
Description: Satisfaction with hospital discharge is measured by the Hospital Consumer Assessment of Healthcare Providers Survey (HCAHPS); "Child HCAHPS" which includes 8 items (range 0-100 with higher values representing higher satisfaction). Response options are "Yes, definitely," "Yes, somewhat" and "No." The items ask about the child and the hospital related to their recent stay.
Time Frame: 7 days post discharge from the hospital
Population: Caregivers who completed the satisfaction measure at the 1 week follow up are included in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care + Intervention (Case) | Usual Care (Control)
Number analyzed (Participants) | 258 | 262
units on a scale | 81.9 (24.8) | 84.2 (23.8)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Usual Care + Intervention (Case) | Usual Care (Control)
All-Cause Mortality (participants affected / at risk) | 0/318 | 0/319
Serious Adverse Events (participants affected / at risk) | 0/318 | 0/319
Other Adverse Events (participants affected / at risk) | 0/318 | 0/319

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04171999/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT04171999/SAP_001.pdf
  • Informed Consent Form (2022-04-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT04171999/ICF_002.pdf